CLINICAL TRIAL: NCT01722227
Title: Anti-diabetic Effects of Liraglutide in Adolescents and Young Subjects With Type 1 Diabetes
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No Funding Received from ADA
Sponsor: University at Buffalo (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Paresh Dandona, Distinguished Professor of Medicine, Kaleida Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1964 Liraglutide ADA; 1-12-CT-20 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide 0.6mg (Active Comparator): Daily Injection
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Daily Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide
  Arms: Liraglutide 0.6mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is the first prospective randomized double-blind placebo-controlled study to investigate the effect of a GLP-1 analog, specifically liraglutide, on blood glucose levels and variability in subjects with type 1 diabetes treated with insulin. Liraglutide is the preferred GLP-1 analog for this study because the pharmacokinetics and pharmacodynamics of the drug are consistent with a sustained duration of action. The current gold standard for management of type 1 diabetes is based on insulin replacement with novel analogs with specified pharmacodynamic profiles or with unique insulin delivery systems (insulin pump therapy). No other adjuvant therapy has demonstrated sustained benefit in this population. This study will also investigate the effect of liraglutide on suppression of glucagon secretion during meal challenges. This is of particular importance since, in the absence of insulin secretion from the β-cell, there is no paracrine inhibition of glucagon secretion by the α-cell. Dysregulation of glucagon secretion may impact the glycemic control and overall pathogenesis in those with type 1 diabetes. The use of CGM technology in this study will allow us to determine the rapidity, consistency, and sustainability of any response to liraglutide.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA:

  1. Females and males with Type 1 diabetes as ascertained by islet autoantibodies (GAD-65 and/or islet cell antibodies)
  2. Age 15-30 years - This age group is being chosen as most will have completed puberty with the accompanying physiologic phase of increased insulin resistance. In addition, this age group shows increased self-management capabilities. Extending the age up to 30 years will allow us to include young adults, since type 1 diabetes is frequently diagnosed in the late teen and early adult years. This study is not powered to detect differences in liraglutide efficacy in different age group but it may provide insight into the effectiveness in the teenage population, in whom optimal glycemic control is often a challenge.
  3. Type 1 diabetes duration greater than 1 year to ensure that a majority of subjects are beyond the partial remission period.
  4. Fasting C-peptide level ≤ 0.3 ng/ml.
  5. HbA1c level equal or less than 9%
  6. Insulin delivery by CSII - the choice is made to facilitate adherence to study drug and also to enable us have a homogeneous group to analyze without having to analyze the data for the covariants of CSII vs. multiple daily injection therapy.
  7. Subjects willing to wear a CGM sensor and perform home blood glucose monitoring four times daily and with symptoms of hypoglycemia.
  8. Subjects well-versed in carbohydrate counting.
  9. BMI < 95th% for age and gender.

Exclusion Criteria:

* EXCLUSION CRITERIA:

  1. Previous exposure to liraglutide
  2. History of abdominal surgery
  3. History of gastroparesis or gastrointestinal reflux disease;
  4. History of acute or chronic pancreatitis
  5. Cirrhosis or hepatic disease defined as transaminases levels > 3 times normal
  6. Impaired renal function defined as serum creatinine >1.5.
  7. HIV or Hepatitis C positive status
  8. Pregnant/breastfeeding females
  9. Individuals with steroid-induced or cystic fibrosis related diabetes
  10. Diabetic Ketoacidosis within 6 months of the study
  11. History of severe hypoglycemia (seizure, loss of consciousness) within 6 months of the study
  12. History of medullary thyroid cancer or MEN2 syndrome
  13. Any other life-threatening cardiac or non-cardiac disease
  14. Participation in a concurrent clinical trial or participation in a trial within 30 days preceding the study period.
  15. Unable to give informed consent/assent.
  16. Adolescents and adults who are considered underweight based on body mass index (BMI):

      1. For adolescents: BMI less than the 5th percentile
      2. For adults: BMI below 18.5

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Mean weekly blood glucose concentrations. | 3 Months
  The primary endpoint of the study is to detect a difference between Liraglutide and placebo groups in the change from baseline in mean weekly blood glucose concentrations after 12 weeks of treatment.

SECONDARY OUTCOMES:
HbA1c | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes-Endocrinology Center of WNY, Williamsville, New York, United States